CLINICAL TRIAL: NCT01704040
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled Study Evaluating CNTO 3157 in Healthy Normal and Asthmatic Subjects Inoculated With Human Rhinovirus Type 16
Brief Title: A Study of CNTO 3157 in Healthy Normal and Asthmatic Participants Inoculated With Human Rhinovirus Type 16
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CR100889; CNTO3157ASH1002 (Other: Janssen Research & Development, LLC); 2011-005369-19 (EudraCT Number)
Record Dates: First submitted 2012-10-08; First posted 2012-10-11 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-12

CONDITIONS: Healthy Volunteers and Asthma
Keywords: Healthy volunteers and asthma; CNTO 3157; Rhinovirus
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Part 1: Healthy participants (CNTO 3157 + HRV-16) (Experimental)
  Interventions: Drug: CNTO 3157 (healthy participants); Other: HRV-16
- Part 1: Healthy participants (placebo + HRV-16) (Placebo Comparator)
  Interventions: Drug: Placebo (healthy participants); Other: HRV-16
- Part 2: Asthmatic patients (CNTO 3157 + HRV-16) (Experimental)
  Interventions: Drug: CNTO 3157 (asthmatic patients); Other: HRV-16
- Part 2: Asthmatic patients (placebo + HRV-16) (Placebo Comparator)
  Interventions: Drug: Placebo (asthmatic patients); Other: HRV-16

INTERVENTIONS:
Drug: CNTO 3157 (healthy participants) — CNTO 3157 10 mg/kg, as a single intravenous infusion, on Day 1, 24 to 72 hours prior to inoculation with human rhinovirus type 16 (HRV-16).
  Arms: Part 1: Healthy participants (CNTO 3157 + HRV-16)
Drug: Placebo (healthy participants) — Placebo, as a single intravenous infusion, on Day 1, 24 to 72 hours prior to inoculation with HRV-16.
  Arms: Part 1: Healthy participants (placebo + HRV-16)
Drug: CNTO 3157 (asthmatic patients) — CNTO 3157 10 mg/kg, as a single intravenous infusion, at Week 1 (Day 1), followed by 3 infusions of 3 mg/kg of CNTO 3157 at Week 2 (Day 8), Week 3 (Day 15), and Week 4 (Day 22). The final infusion (Week 4) will occur 24 to 72 hours prior to inoculation with HRV-16.
  Arms: Part 2: Asthmatic patients (CNTO 3157 + HRV-16)
Drug: Placebo (asthmatic patients) — Placebo, as 4 intravenous infusions, at Week 1 (Day 1), Week 2 (Day 8), Week 3 (Day 15), and Week 4 (Day 22). The final infusion (Week 4) will occur 24 to 72 hours prior to inoculation with HRV-16.
  Arms: Part 2: Asthmatic patients (placebo + HRV-16)
Other: HRV-16 — Single inoculation of HRV-16 in a total volume of approximately 1.0 mL, administered as 2 instillations per naris.

SUMMARY:
The main purposes of this study are to evaluate the safety (Parts 1 and 2) and efficacy (Part 2) of pretreatment with CNTO 3157 in healthy adult and asthmatic adult participants before and after intranasal (into the nose) inoculation with human rhinovirus type 16 (HRV-16).

DETAILED DESCRIPTION:
This is a two-part, randomized (participants are assigned to treatment by chance), double-blind (participants and investigators do not know what study agent is being administered), placebo-controlled study. A placebo appears identical to a study agent, has no active ingredients, and helps investigators evaluate the effect of a study agent. In Part 1, following administration of CNTO 3157 or placebo, the severity of an upper respiratory tract infection, due to inoculation with HRV 16, will be assessed in healthy participants for safety reasons. In Part 2, following administration of CNTO 3157 or placebo and inoculation with HRV-16, efficacy and safety will be assessed in asthmatic participants using standard assessments to evaluate asthma treatments. The study (Parts 1 and 2) will be completed when the last participant completes the last visit (Week 11) in Part 2.

ELIGIBILITY:
Inclusion Criteria:

* Understanding of the study and a signed informed consent form before any study-related procedures
* Willing and able to adhere to the restrictions specified in the protocol
* Results of the following laboratory tests within the following limits: serum alanine aminotransferase (ALT) levels ≤2 x ULN; serum aspartate aminotransferase (AST) levels ≤2 x ULN
* Part 1 (healthy participants):
* a). Body weight in the range of 40 to 125 kg, inclusive. Have a body mass index (BMI) of 19 to 32 kg/m2, inclusive
* b). Healthy with no clinically significant abnormalities as determined by medical history, physical examination, blood chemistry assessments, hematologic assessments, coagulation and urinalysis, measurement of vital signs, and 12-lead electrocardiogram (ECG) performed at Screening Visit 2
* Part 2:
* a). (BMI) of 19 to 40 kg/m2, inclusive; have a physician-documented diagnosis of asthma for at least 6 months prior to Screening Visit 2; have stable asthma based on physician assessment at Screening Visit 2
* b). Have an Asthma Control Questionnaire (ACQ) symptom score less than (<)2.5 at Screening Visit 2
* c). Have a prebronchodilator forced expiratory volume in the first second (FEV1) greater than or equal to (>=) 65 percent of predicted normal value at Screening Visit 2

Exclusion Criteria:

* Part 1 (healthy participants): Has any condition that in the opinion of the investigators, would constitute a risk or a contraindication for participating in the study, prevent the participant from meeting or performing study requirements, or could interfere with the study objectives, conduct, or evaluation
* At Screening Visit 1 and throughout the study, works with (or lives with a family member who cares for) the elderly, (eg, nursing home), or lives with someone who may be at risk from transmission of the human rhinovirus type 16 (HRV-16) challenge agent, including, but not limited to, individuals with chronic lung disease (including asthma), a premature infant, or an immunocompromised individual
* Has had any acute illness, including a common cold, within 4 weeks prior to Screening Visit 1, or has had a major illness or hospitalization within 6 months prior to Screening Visit 1
* Has active allergic rhinitis or perennial allergy symptoms (eg, due to ragweed) at Screening Visit 2 or expects to have active allergic rhinitis or perennial allergy symptoms during the study
* Has a current infection (eg, sepsis, pneumonia or pyelonephritis), or has been hospitalized and/or received antimicrobials for a serious infection during the 6 months prior to Screening Visit 1
* Part 2 (asthmatic patients): Has a history of any other chronic lung disease, including chronic obstructive pulmonary disease (COPD), bronchiolitis, bronchiectasis, allergic bronchopulmonary aspergillosis (mycosis), occupational asthma, sleep apnea, pulmonary hypertension, or any other obstructive pulmonary disease, liver or renal insufficiency; significant unstable cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances, or other body system disorders that are clinically significant in the opinion of the investigator
* Has ever had an episode of life-threatening asthma defined as respiratory arrest or requiring intubation for asthma
* Has been hospitalized (for greater than 24 hours) due to asthma in the 5 years prior to Screening Visit 1
* Has experienced an asthma exacerbation in the 12 weeks prior to Screening Visit 1 requiring management with systemic steroids
* Is receiving a high-dose inhaled corticosteroid (ICS) (>500 µg/day to fluticasone or equivalent). Use of low or medium dose ICS (≤500 µg/day fluticasone or equivalent) with or without permitted controller medications, eg, long-acting Beta2 agonists (LABA), leukotriene receptor antagonists (LTRA), is allowed

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2012-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
The maximum percent decrease relative to baseline in the prebronchodilator forced expiratory volume in 1 second (FEV1) measurements (Part 2) | Up to 10 days after inoculation with human rhinovirus type 16 (HRV-16)

SECONDARY OUTCOMES:
Area under the serum concentration versus time curve (AUC) of change from baseline in Cold Symptom Assessment Score | Up to 10 days after inoculation with HRV-16
  Cold symptoms is rated using a 5 point scale (0=none and 4=very severe). Scores can range from 0-32, with higher scores indicating more symptoms.
AUC of change from baseline in Cold and Chest Symptom Scale | Up to 10 days after inoculation with HRV-16
  Cold and chest symptoms are rated using a 5 point scale: 0 using a 5 point scale (0=none and 4=very severe). Scores can range from 0-60, with higher scores indicating more symptoms.
AUC of change from baseline in log-transformed fractional concentration of exhaled nitric oxide (FENO) | Up to 10 days after inoculation with HRV-16
AUC of the percent change from baseline in clinic assessed prebronchodilator FEV1 | Up to 10 days after inoculation with HRV-16
AUC of change from baseline in morning (AM) peak expiratory flow rate (PEFR) | Up to 10 days after inoculation with HRV-16
AUC of the change from baseline in prebronchodilator percent predicted FEV1 | Up to 10 days after inoculation with HRV-16
AUC of the change from baseline in prebronchodilator forced vital capacity (FVC) | Up to 10 days after inoculation with HRV-16
AUC of the change from baseline in prebronchodilator forced expiratory flow at 25 to 75% of vital capacity (FEV25-75) | Up to 10 days after inoculation with HRV-16
AUC of the change from baseline in prebronchodilator FEV1/FVC | Up to 10 days after inoculation with HRV-16
AUC of change from baseline in average total asthma symptom diary score | Up to 10 days after inoculation with HRV-16
Change from baseline in Asthma Control Questionnaire (ACQ) | Up to 10 days after inoculation with HRV-16
  ACQ is an instrument designed to evaluate asthma control. Seven items are scored on a 7-point scale (0=good control, 6=poor control) with the mean score as an overall summary score. Questions 1-6 are completed by the patient; the last item is entered by site personnel and corresponds to the patient's percent predicted FEV1 categorized according to the 7-point scale. Higher scores reflect poorer control.
Change from baseline in Cold Symptom Assessment Score | Up to 11 weeks
  Clinical symptoms to HRV-16 will be assessed by using the Cold Symptom Assessment Score, wherein participants will report the presence and severity of their cold symptoms in the context of the previous 24 hours via an interactive interview with the study staff. The symptoms consist of nasal congestion (stuffy nose), rhinorrhea (runny nose), sore throat, sneezing, cough, headache, malaise (feeling run down, tired) and chilliness. Severity is rated using a 5 point scale (0=none, 1=mild, 2=moderate, 3=severe, and 4=very severe). Scores can range from 0-32, with higher scores indicating more symptoms.
Change from baseline in Cold and Chest Symptom Scale | Up to 11 weeks
  The Cold and Chest Symptom Scale contains 15 items composing 2 domains, a total cold score and a total chest score. Together, these 2 domains comprise the chest symptom assessment score.
  Total Cold Score domain: sneezing, runny nose, blocked or stuff nose, sore throat or hoarse voice, headache or face pain, generally unwell, chills, fever or shivery and cough and Total Chest Score domain: cough on waking, wheeze on waking, daytime cough, daytime wheeze, daytime chest tightness, daytime breathlessness and nocturnal cough, wheeze and breathlessness.
  Severity is rated using a 5 point scale: 0 using a 5 point scale (0=none, 1=mild, 2=moderate, 3=severe, and 4=very severe). Scores can range from 0-60, with higher scores indicating more symptoms.
Change from baseline in log-transformed FENO over time | Up to 11 weeks
Change from baseline over time in prebronchodilator and postbronchodilator FEV1 | Up to 11 weeks
Change from baseline over time in percent-predicted prebronchodilator and postbronchodilator FEV1 | Up to 11 weeks
Change from baseline over time in prebronchodilator and postbronchodilator FVC | Up to 11 weeks
Change from baseline over time in prebronchodilator and postbronchodilator FEV25-75 | Up to 11 weeks
Change from baseline over time in prebronchodilator and postbronchodilator FEV1/FVC | Up to 11 weeks
Change from baseline in morning/evening PEFR over time | Up to 11 weeks
Change from baseline in Total Nasal and Ocular Symptom Score (TNOSS) | Up to Day 22
  Nose and eye symptoms are rated by the patient using a 5-point categorical response scale from 0 to 4, where 0 indicates absent/no symptom, and 4 indicates extremely severe symptoms, with a 24-hour recall period.
Change from baseline in average total asthma symptom diary score | Up to 11 weeks
Change from baseline in average number of nocturnal awakenings | Up to 11 weeks
Change from baseline in average rescue medication use over time | Up to 11 weeks
Number of symptom-free days | Up to 10 days after inoculation with HRV-16
The maximum decrease from baseline in the prebronchodilator FEV1 measurements | Up to 10 days after inoculation with HRV-16
Time to the maximum decrease relative to baseline in prebronchodilator FEV1 | Up to 10 days after inoculation with HRV-16

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (13):
- Antwerp, Belgium
- Canada (2):
  - Calgary, Alberta
  - Halifax, Nova Scotia
- Denmark (2):
  - Hellerup
  - København NV
- Germany (2):
  - Borstel
  - Frankfurt
- Netherlands (2):
  - Amsterdam-Zuidoost
  - Groningen
- United Kingdom (4):
  - Belfast
  - Dundee
  - London
  - Manchester

REFERENCES:
- [Derived] Silkoff PE, Flavin S, Gordon R, Loza MJ, Sterk PJ, Lutter R, Diamant Z, Turner RB, Lipworth BJ, Proud D, Singh D, Eich A, Backer V, Gern JE, Herzmann C, Halperin SA, Mensinga TT, Del Vecchio AM, Branigan P, San Mateo L, Baribaud F, Barnathan ES, Johnston SL. Toll-like receptor 3 blockade in rhinovirus-induced experimental asthma exacerbations: A randomized controlled study. J Allergy Clin Immunol. 2018 Apr;141(4):1220-1230. doi: 10.1016/j.jaci.2017.06.027. Epub 2017 Jul 20. PMID 28734844